CLINICAL TRIAL: NCT06942780
Title: Preliminary Efficacy and Feasibility Analysis of Cognitive Training, Group Social Activities, Physical Exercise, and MIND Diet in Patients With Mild Cognitive Impairment
Brief Title: Evaluation of the Effect of Healthy Lifestyle Intervention for Patients With Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202504
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: Cognitive training; MIND diet; social; exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Social Work; Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the usual care group (Sham Comparator): The usual care group was given a health education booklet on the importance of proper diet, physical activity, cognitive exercise, and social interaction to help participants establish a basic understanding of these healthy lifestyles and try to do them. The manual teaches about common healthy ingredients, the appropriate frequency and intensity of aerobic exercise, and the benefits of brain games, reading, and learning new skills. And specific forms of social communication, such as participation in community activities, regular gatherings with relatives and friends.
  Interventions: Behavioral: Health Education Manual
- the comprehensive intervention group (Active Comparator): The intervention measures of the comprehensive intervention group were divided into exercise intervention, group socializing, MIND diet education and cognitive training. Twice a week for eight weeks.
  Interventions: Behavioral: Exercise intervention; Behavioral: Social intervention; Behavioral: Dietary intervention; Behavioral: Cognitive intervention; Behavioral: Health Education Manual

INTERVENTIONS:
Behavioral: Exercise intervention — The multi-component exercise mode is adopted, and the three-stage structured design of "warm-up preparation - main training - finishing and relaxation" is adopted, and the participants' heart rate is monitored in real time with the exercise bracelet throughout the whole process to ensure that the training intensity is reached. The movement process is guided synchronously by the video music teaching system, and the specific process is as follows:
  1. Warm-up preparation (3 minutes) : Warm up the head and neck, shoulder joints, arms and wrists, waist and abdomen, thighs and ankles in turn, and perform 30 seconds for each movement.
  2. Main training stage (60min) : aerobic exercise adopts basic steps of square dance or advanced step training; The resistance training module carries out compound resistance exercises of sitting posture, leg lift and arms forward lift.
  3. Finishing and relaxing stage (12min) : select the traditional health exercise eight Duan Jin.
  Arms: the comprehensive intervention group
Behavioral: Social intervention — The duration of each intervention was 40min, mainly group social interaction, guided by professionals (medical social workers). Divided into three stages:
  The first stage (3min) : The facilitator will go through small jokes, soothing music, etc.Create a relaxed atmosphere and briefly introduce the theme of the week.
  The second stage (35min) : During the activity, participants began to chat around the theme, and the host guided them timely.
  The third stage (2min) : Summarize the intervention and praise the participants.
  Arms: the comprehensive intervention group
Behavioral: Dietary intervention — The researcher distributed the health education manual of the cognitive disorder diagnosis and treatment center, and conducted a 5-minute MIND diet health education, explaining relevant dietary requirements and focusing on the collocation of one type of food every week. The participants were then given homework that asked them to strictly follow the MIND diet in their daily diet. At the same time, the participants' caregivers are required to upload photos of their daily meals to the wechat group for supervision and feedback.
  Arms: the comprehensive intervention group
Behavioral: Cognitive intervention — Cognitive digital therapy was adopted, and participants were supervised by their caregivers for 5 days a week and 30min each time for cloud-based home training (avoiding 2 hospital intervention days) for 8 weeks. The training covers core cognitive functions such as attention, memory and logical reasoning.
  Arms: the comprehensive intervention group
Behavioral: Health Education Manual — Distribute health education handbooks to guide patients to establish a good awareness of a healthy lifestyle. The manual can popularize health knowledge, covering various aspects such as diet, exercise, and rest, enabling patients to understand the importance of a healthy lifestyle, encouraging them to actively improve their living habits, slow down the progression of the disease, and enhance their quality of life.

SUMMARY:
This clinical study aims to evaluate the feasibility and preliminary effectiveness of a comprehensive lifestyle intervention program for patients with mild cognitive impairment. The intervention consists of four components: cognitive training, physical exercise, MIND diet, and group social activities.

The hypothesis is that this integrated healthy lifestyle intervention may slow cognitive decline, improve daily functional abilities, and enhance the quality of life in MCI patients. Feasibility will be assessed based on participation rates, program completion rates, and participant satisfaction. Effectiveness will be evaluated using scales such as MoCA, MMSE.

The study participants will be clinically diagnosed mild cognitive impairment patients. If feasibility is confirmed, the results will provide a basis for larger-scale clinical trials and offer insights into non-pharmacological intervention strategies for brain health in high-risk populations.

DETAILED DESCRIPTION:
Research Background

1. MCI Status and Impact Mild Cognitive Impairment (MCI) is an intermediate state between normal aging and dementia, characterized by cognitive decline. Globally, the prevalence of MCI among individuals aged 65 and older is approximately 15%-20%, while in China, the prevalence among those aged 60 and older is 15.5%, affecting approximately 38.77 million people.

   MCI patients experience cognitive decline, reduced quality of life, and increased economic burden on families (approximately 20%-30% higher than healthy elderly individuals). The prevalence of depressive symptoms in MCI patients is significantly higher than in healthy elderly individuals.

   MCI patients have a high risk of progressing to dementia, with an annual conversion rate of 10%-15%, and up to 50% progressing within five years. However, early intervention can reverse or delay the progression to dementia.
2. Importance of Healthy Lifestyle Interventions. A healthy lifestyle, including observable behaviors (e.g., diet, exercise) and indirect behaviors (e.g., psychological state, cognitive ability), plays a significant role in preventing and intervening in MCI.

   Exercise Intervention: Regular exercise (e.g., brisk walking, resistance training, Tai Chi) improves cognitive function. It is recommended that older adults with cognitive decline engage in 150-300 minutes of moderate-intensity activity per week.

   Social Intervention: Active social participation (e.g., interest groups, health education) reduces the risk of cognitive decline. It is recommended that MCI patients participate in social activities at least twice a week.

   Dietary Intervention: The MIND diet (a combination of the Mediterranean and DASH diets) emphasizes antioxidant and anti-inflammatory foods, reducing MCI risk and slowing age-related cognitive decline.

   Cognitive Intervention: Cognitive training (e.g., digital cognitive therapy) is effective in improving intervention outcomes. It is recommended that MCI patients undergo at least 3 sessions per week, each lasting 30 minutes, with a total training time of no less than 20 hours.
3. Research Status and Significance Current research on healthy lifestyle interventions for MCI patients is limited, with most studies focusing on single interventions rather than comprehensive approaches.

This study combines exercise, social activities, diet, and cognitive training to systematically evaluate the comprehensive effects of multidimensional healthy lifestyle interventions. The findings will provide evidence for developing personalized and precise intervention strategies, helping to reduce the risk of dementia conversion, alleviate family and societal burdens, and promote healthy aging.

Statistical Methods The SPSS 23.0 statistical software was used to build the database and conduct statistical analyses. Descriptive statistics were applied to describe the basic characteristics of the study subjects and the outcome indicators of the feasibility analysis. For measurement data, the Shapiro-Wilk test was used to test for normality. Normally distributed data were described using means and standard deviations, while non-normally distributed data were described using medians and interquartile ranges. Categorical data were described using frequencies and percentages.

For the outcome indicators of the effectiveness validation of the study subjects, between-group differences were analyzed. Normally distributed data were analyzed using the independent samples t-test, while non-normally distributed data were analyzed using the Mann-Whitney U test. A two-tailed p-value ≤0.05 was considered statistically significant.

Innovations

1. Perspective Innovation Starting from an overall healthy lifestyle and focusing on MCI patients, this study integrates multi-factorial interventions (exercise, diet, social interaction, and cognitive training), breaking the limitations of traditional single-factor research. Meanwhile, the intervention effects are evaluated from multiple dimensions to comprehensively measure the impact of lifestyle interventions on MCI patients.
2. Methodological Innovation Combining multi-modal interventions (cognitive training, exercise, MIND diet, group social activities) with digital technology (cognitive digital therapy, fitness trackers for heart rate monitoring), this study enables real-time multi-dimensional monitoring and data collection, enhancing intervention compliance and engagement.
3. Application Innovation Focusing on modifiable factors in the lives of MCI patients, this study designs practical interventions that can be implemented in both family and community settings. Based on the research findings, an integrated promotion model of "hospital-community-family" can be established to effectively improve the accessibility and sustainability of the interventions.
4. Research Framework Innovation This study constructs a comprehensive intervention framework that integrates diet, exercise, cognition, and social interaction, providing a reference for future research.

ELIGIBILITY:
Inclusion Criteria:

1. To meet the diagnostic criteria of MCI, refer to the diagnostic criteria of MCI in "2018 Chinese Guidelines for the Diagnosis and Treatment of Dementia and Cognitive Impairment (5) : Diagnosis and Treatment of Mild Cognitive Impairment".
2. Have caregiver > 6 months.
3. Participate in the study voluntarily and sign the informed consent.

Exclusion Criteria:

1. Have received other cognitive intervention therapy recently (within 6 months).
2. Diagnosis of functional encephalopathy or obvious mental disorders, such as Parkinson's disease, epilepsy, schizophrenia.
3. Suffering from serious cardiovascular diseases, malignant tumors and other major physical diseases.
4. Have visual, hearing, speech or limb dysfunction, unable to complete the test.
5. Patients with chronic diseases who have special dietary needs or require special dietary management.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Participation rate | Baseline
  Recruitment success rate : number of people who agree to participate/total number of people eligible and invited
Study Measures Completion | 4 weeks and 8weeks
  Number of participants with full protocol compliance, including: attending interventions as scheduled, verifying target exercise intensity via fitness trackers, and recording MIND diet adherence in the WeChat group.
Montreal Cognitive Assessment | Baseline and 8 weeks
  Seven sub-dimensions, including visuospatial/executive function, naming, attention, language, abstract ability, delayed recall and orientation, were scored out of 30, with higher scores indicating better cognitive ability. The sensitivity and specificity of the Beijing version of MoCA scale were 0.92, 0.84, 0.86, and 0.82 Cronbach'sa coefficient of internal consistency.
Mini-Mental State Examination | Baseline and 8 weeks
  The scale includes the assessment of orientation, attention and computing ability, immediate recall, delayed recall, language function and visuospatial ability. The total score is 30 points, the higher the score is, the better the cognitive function, >27 is normal, <27 is cognitive dysfunction. The Chinese MMSE retest reliability is 0.90.

SECONDARY OUTCOMES:
12-item Short-Form Health Survey | Baseline and 8 weeks
  The total score of the scale ranges from 12 to 65 points. The higher the scale score, the better the quality of life. When the 12-item Short-Form Health Survey was applied to the elderly population in China, the Cronbach'sa coefficient of the scale was 0.775, indicating good reliability and validity.
Social Support Rating Scale | Baseline and 8 weeks
  The scale consisted of 10 items and 3 dimensions (subjective support, objective support and utilization of social support), with a total score of 12 to 66 points, and the higher the score, the better the social support. The retest reliability of the scale was 0.92, and the prediction validity was good.
Geriatric Depression Scale | Baseline and 8 weeks
  Geriatric Depression Scale is adapted by Sheikh and other scholars on the basis of the standard edition, with a total of 15 items, each item is 1 point. The scale scores range from 0 to 15 points. The higher the score, the more likely it is to have depressive symptoms. The Chinese version of GDS-15 scale has good applicability in the elderly population in China, with a one-week retest reliability of 0.728 and a Cronbach'sa coefficient of 0.793.
General information questionnaire | Baseline
  demographic information (age, sex, education, marital status, etc.), health status (medical history, drug use, smoking and alcohol use), lifestyle (physical activity, eating habits, social activities).
Satisfaction Questionnaire | 8weeks
  The satisfaction questionnaire covers four aspects (cognitive training, exercise, MIND diet and social activities), and gives the scores of acceptability (interest/difficulty), time commitment and overall satisfaction (5-point Likert scale), with a total score ranging from 13 to 65 points. The higher the score is, the more satisfied one will be. Open-ended questions will collect suggestions for improvement.
Occurrence of adverse events | From enrollment to the end of the intervention at eight weeks
  The number of cases of falls and muscle injuries during exercise, indigestion and gastrointestinal reactions caused by following the MIND diet

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data Sensitivity: Cognitive health datasets contain detailed personal health and lifestyle information that, even anonymized, could carry re-identification risks for vulnerable populations like older adults.
  Resource Limitations: Our team currently lacks dedicated infrastructure to responsibly anonymize, curate, and manage external data requests while ensuring compliance with evolving data protection laws.

REFERENCES:
- [Background] Zhang Lixiu, Liu Xueqin. Study on the reliability and validity of the Chinese version of the Montreal Cognitive Assessment Scale J. Nursing Research, 2007, (31): 2906-7.
- [Background] The theoretical basis and research application of Social Support Rating Scale J. Journal of Clinical Psychiatry, 1994, (02): 98-100.
- [Background] Zhou Xiaoxuan, Xie Min, Tao Jing, et al. Research and application of simple intelligent mental state examination scale J. Chinese Journal of Rehabilitation Medicine, 2016, 31(06): 694-696.
- [Background] Mitchell AJ, Bird V, Rizzo M, Meader N. Diagnostic validity and added value of the Geriatric Depression Scale for depression in primary care: a meta-analysis of GDS30 and GDS15. J Affect Disord. 2010 Sep;125(1-3):10-7. doi: 10.1016/j.jad.2009.08.019. Epub 2009 Oct 2. PMID 19800132
- [Background] Sheikh J. Geriatric depression scale (GDS): recent evidence and development of ashorter version J. Clin Gerontol, 1986, 5(1): 165-173.
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Lu L, Cai S, Xiao Q, Peng J, Li F, Li Y, Li B, Li T, Rong S. The association between Chinese adapted MIND diet and cognitive function in Chinese middle-aged and older adults: results from the Chinese Square Dance Cohort. Eur J Nutr. 2024 Nov 23;64(1):22. doi: 10.1007/s00394-024-03522-8. PMID 39579171
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] van den Brink AC, Brouwer-Brolsma EM, Berendsen AAM, van de Rest O. The Mediterranean, Dietary Approaches to Stop Hypertension (DASH), and Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diets Are Associated with Less Cognitive Decline and a Lower Risk of Alzheimer's Disease-A Review. Adv Nutr. 2019 Nov 1;10(6):1040-1065. doi: 10.1093/advances/nmz054. PMID 31209456
- [Background] Chinese Expert Consensus Committee on Brain and Cognitive Health Management, Editorial Committee of Chinese Journal of Health Management. Chinese expert consensus on brain cognitive health management (2023) J. Chinese Journal of Health Management, 2023, 17(12): 881-892.
- [Background] Special Committee of Neurodegeneration, Chinese Society of Microcirculation, Neuropsychological and Behavioral Neurology Group, Chinese Society of Neurology, Neurorehabilitation Group, Chinese Society of Neurology. Chinese expert consensus on rehabilitation management of Alzheimer's disease J. Chinese Journal of Gerontology, 2020, 39(1): 9 19.
- [Background] Expert group on Exercise Prescription in China Expert Consensus (2023). Chinese expert consensus on exercise prescription (2023) J. Chinese Journal of Sports Medicine, 2023, 42(1): 3 13.
- [Background] Chinese Geriatrics Society. [Chinese expert consensus on multidisciplinary decision-making model for mobility limitation in older adults (2024 edition)]. Zhonghua Yi Xue Za Zhi. 2024 Mar 26;104(12):893-905. doi: 10.3760/cma.j.cn112137-20230816-00238. Chinese. PMID 38514338
- [Background] China Geriatric Nursing Alliance, Xiangya Nursing School of Central South University (Xiangya Pan-Sea Health Management Research Institute of Central South University), Xiangya Hospital of Central South University (National Clinical Medical Research Center for Geriatric Diseases), etc. Clinical practice guidelines for non-drug intervention in the elderly with cognitive decline: Physical activity J. Chinese Journal of General Medicine, 2023, 26(16): 1927-1937+1971.
- [Background] Committee for the preparation of Physical Activity Guidelines for Chinese People. Physical activity guidelines for Chinese population (2021) J. Chinese Journal of Epidemiology, 2022, 43(1): 56.
- [Background] American College of Sports Medicine; Chodzko-Zajko WJ, Proctor DN, Fiatarone Singh MA, Minson CT, Nigg CR, Salem GJ, Skinner JS. American College of Sports Medicine position stand. Exercise and physical activity for older adults. Med Sci Sports Exerc. 2009 Jul;41(7):1510-30. doi: 10.1249/MSS.0b013e3181a0c95c. PMID 19516148
- [Background] Hsu CL, Best JR, Davis JC, Nagamatsu LS, Wang S, Boyd LA, Hsiung GR, Voss MW, Eng JJ, Liu-Ambrose T. Aerobic exercise promotes executive functions and impacts functional neural activity among older adults with vascular cognitive impairment. Br J Sports Med. 2018 Feb;52(3):184-191. doi: 10.1136/bjsports-2016-096846. Epub 2017 Apr 21. PMID 28432077
- [Background] McMaster M, Kim S, Clare L, Torres SJ, D'Este C, Anstey KJ. Body, Brain, Life for Cognitive Decline (BBL-CD): protocol for a multidomain dementia risk reduction randomized controlled trial for subjective cognitive decline and mild cognitive impairment. Clin Interv Aging. 2018 Nov 21;13:2397-2406. doi: 10.2147/CIA.S182046. eCollection 2018. PMID 30538436
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Zhao QF, Tan L, Wang HF, Jiang T, Tan MS, Tan L, Xu W, Li JQ, Wang J, Lai TJ, Yu JT. The prevalence of neuropsychiatric symptoms in Alzheimer's disease: Systematic review and meta-analysis. J Affect Disord. 2016 Jan 15;190:264-271. doi: 10.1016/j.jad.2015.09.069. Epub 2015 Oct 24. PMID 26540080
- [Background] Jia L, Du Y, Chu L, Zhang Z, Li F, Lyu D, Li Y, Li Y, Zhu M, Jiao H, Song Y, Shi Y, Zhang H, Gong M, Wei C, Tang Y, Fang B, Guo D, Wang F, Zhou A, Chu C, Zuo X, Yu Y, Yuan Q, Wang W, Li F, Shi S, Yang H, Zhou C, Liao Z, Lv Y, Li Y, Kan M, Zhao H, Wang S, Yang S, Li H, Liu Z, Wang Q, Qin W, Jia J; COAST Group. Prevalence, risk factors, and management of dementia and mild cognitive impairment in adults aged 60 years or older in China: a cross-sectional study. Lancet Public Health. 2020 Dec;5(12):e661-e671. doi: 10.1016/S2468-2667(20)30185-7. PMID 33271079
- [Background] Li X, Feng X, Sun X, Hou N, Han F, Liu Y. Global, regional, and national burden of Alzheimer's disease and other dementias, 1990-2019. Front Aging Neurosci. 2022 Oct 10;14:937486. doi: 10.3389/fnagi.2022.937486. eCollection 2022. PMID 36299608